CLINICAL TRIAL: NCT05662930
Title: Diyabetik Hipertansif Hastalarda Stres Yanıtının Değerlendirilmesi
Brief Title: Evaluation Of Stress Response In Diabetic Hypertensive Patients
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Iliriana Alloqi Tahirbegolli, Principal investigator, Istanbul University
Other Study IDs: 22939
Record Dates: First submitted 2022-08-01; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Diabetes; Hypertension
Keywords: Diabetes mellitus; Hypertension; Cortisol; Stress; Aldosterone
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypertension + Diabetes Mellitus (HT+DM): Patients who fulfilled the following criteria were included in this group:
  1. Using antihypertensive treatment for the last 3 months
  2. Diagnosed with Type 2 Diabetes Mellitus and taking medication for at least 3 months
  3. Being between the ages of 40-65
  4. Being male
  5. Having signed the informed consent form
  Interventions: Behavioral: First arithmetic problem solving; Behavioral: Second arithmetic problem solving; Behavioral: Third arithmetic problem solving; Behavioral: Fourth arithmetic problem solving; Behavioral: Fifth arithmetic problem solving; Behavioral: Sixth arithmetic problem solving
- Hypertension (HT): Patients who fulfilled the following criteria were included in this group:
  1. Using antihypertensive treatment for the last 3 months
  2. Being between the ages of 40-65
  3. Being male
  4. Having signed the informed consent form
  Interventions: Behavioral: First arithmetic problem solving; Behavioral: Second arithmetic problem solving; Behavioral: Third arithmetic problem solving; Behavioral: Fourth arithmetic problem solving; Behavioral: Fifth arithmetic problem solving; Behavioral: Sixth arithmetic problem solving

INTERVENTIONS:
Behavioral: First arithmetic problem solving — In a quiet environment, a white paper in A4 format was placed in front of the patient on the table, and the patients were asked to subtract the number 3 from 2907 for 100 seconds.
  The researcher was standing in front of the patient and asks to make corrections by giving a warning whenever the patient made a mistake in the calculation.
Behavioral: Second arithmetic problem solving — In the same A4-sized white paper that was placed in front of each patient on a table, immediately after the first subtraction process, patients were asked to subtract 7 from 6828 for another 100 seconds.
  When the patient made a calculating error, the researcher stood in front of the patient and asked them to make corrections by issuing a warning.
Behavioral: Third arithmetic problem solving — In the same A4-sized white paper that was placed in front of each patient on a table, immediately after the previous subtraction process, patients were asked to subtract 13 from 9561 for another 100 seconds.
  When the patient made a calculating error, the researcher stood in front of the patient and asked them to make corrections by issuing a warning.
Behavioral: Fourth arithmetic problem solving — In the same A4-sized white paper that was placed in front of each patient on a table, immediately after the previous subtraction process, patients were asked to subtract 8 from 5113 for another 100 seconds.
  When the patient made a calculating error, the researcher stood in front of the patient and asked them to make corrections by issuing a warning.
Behavioral: Fifth arithmetic problem solving — In the same A4-sized white paper that was placed in front of each patient on a table, immediately after the previous subtraction process, patients were asked to subtract 14 from 8318 for another 100 seconds.
  When the patient made a calculating error, the researcher stood in front of the patient and asked them to make corrections by issuing a warning.
Behavioral: Sixth arithmetic problem solving — In the same A4-sized white paper that was placed in front of each patient on a table, immediately after the previous subtraction process, patients were asked to subtract 17 from 9994 for another 100 seconds.
  When the patient made a calculating error, the researcher stood in front of the patient and asked them to make corrections by issuing a warning.

SUMMARY:
In this research, we aimed to examine salivary cortisol changes in the cognitive stress response of patients with Hypertension + Diabetes Mellitus (HT+DM) and Hypertension (HT) and to determine the differences between them.

The research was conducted by solving an arithmetic task as a stress test in 62 patients with HT+DM and HT that are being treated in the outpatient clinic of Medical Pharmacology and Clinical Pharmacology Department at Istanbul University, Istanbul Medical Faculty Hospital.

DETAILED DESCRIPTION:
In this study, saliva samples were taken for cortisol measurement, and patients were instructed to place the cotton piece in the salivette® tubes directly into their mouths without touching it with anything, hold it for 30-60 seconds, and then insert it back into the tubes in the same way, four times total, once before arithmetic stress and three times after stress, on Tuesdays, Wednesdays, and Thursdays between the hours of 12:00-16:00.

Salivary cortisol was measured using the electro-chemiluminescence immunoassay.

ELIGIBILITY:
Inclusion Criteria:

1. Using antihypertensive treatment for the last 3 months
2. Diagnosed with Type 2 Diabetes Mellitus and taking medication for at least 3 months
3. Being between the ages of 40-65
4. Being male
5. Having signed the informed consent form

Exclusion Criteria:

1. Female gender
2. Patients younger than 40 years old or older than 65 years old
3. Uncontrolled blood pressure (SBP>140 mmHg, DBP>90 mmHg)
4. Using antipsychotic medication
5. Using current treatment for less than 3 months
6. Having a previous MI
7. Having a previous stroke
8. Having a lung disease
9. Having organ failure
10. Having Cushing's disease
11. Having aldosteronism
12. Failure to sign the informed consent form

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants were male based on self-representation of gender identity.
Study Population: The study population consisted of patients in the register of the pharmacology clinic of the faculty of medicine who have a diagnosis of hypertension and diabetes mellitus type 2.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Cortisol | Baseline
  A saliva sample is collected for cortisol evaluation
Cortisol | 30 minutes after beginning
  A saliva sample is collected
Cortisol | 45 minutes after beginning
  A saliva sample is collected
Cortisol | 60 minutes after beginning
  A saliva sample is collected
Blood pressure | Baseline
  The patient is rested by sitting before the measurement
Blood pressure | 15 minutes after beginning measurement
  The patient is rested by sitting before the measurement
Blood pressure | 35 minutes after beginning measurement
  The patient is rested by sitting before the measurement
Blood pressure | 50 minutes after beginning measurement
  The patient is rested by sitting before the measurement
Blood pressure | 75 minutes after beginning measurement
  The patient is rested by sitting before the measurement
Aldosterone | Baseline
  Venous blood sample is collected
Heart Rate | Beginning
  The patient is rested by sitting before the measurement
Heart Rate | 15 minutes after beginning
  The patient is rested by sitting before the measurement
Heart Rate | 35 minutes after beginning
  The patient is rested by sitting before the measurement
Heart Rate | 50 minutes after beginning
  The patient is rested by sitting before the measurement
Heart Rate | 75 minutes after beginning
  The patient is rested by sitting before the measurement

SECONDARY OUTCOMES:
Mental state examination | Baseline
  Mini Mental State Examination - MMSE is used to evaluate the mental state
Physical activity | Baseline
  International Physical Activity Questionnaire is used to evaluate the level of physical activity
Health related Quality of life | Baseline
  SF-36 v2 is used to evaluate the health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Iliriana Alloqi Tahirbegolli, Prof.Ass.Dr., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Based on the regulations it is not mandatory for this study to share the individual data of patients. But in the case of a proper request by researchers the data can be shared by the principal researcher of the study.

REFERENCES:
- [Derived] Alloqi Tahirbegolli I, Tahirbegolli B, Sen S, Sayin B, Kaskal M, Uresin AY. Evaluation of Stress Response in Middle-Aged Male Diabetic Hypertensive Patients. J Clin Endocrinol Metab. 2023 Aug 18;108(9):2307-2314. doi: 10.1210/clinem/dgad122. PMID 36880261